CLINICAL TRIAL: NCT06278051
Title: Post-Marketing Database Study for Rivaroxaban in Patients With Pediatric VTE
Brief Title: An Observational Study to Learn More About How Safe Treatment With Rivaroxaban is in Children in Japan With Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Pharmaceutical Companies (formerly Johnson & Johnson Pharmaceutical Research & Development L.L.C.) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21411
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Suspensions; Rivaroxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Xarelto (Rivaroxaban, BAY59-7939)
  Interventions: Drug: Rivaroxaban granules for oral suspension
- Warfarin
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban granules for oral suspension — Treatment dose and period decided by its prescription
  Other Names: Xarelto, BAY59-7939
  Groups: Xarelto (Rivaroxaban, BAY59-7939)
Drug: Warfarin — Treatment dose and period decided by its prescription
  Groups: Warfarin

SUMMARY:
This is an observational study in which only data will be collected from children with venous thromboembolism who are prescribed rivaroxaban or warfarin by their doctors.

Venous thromboembolism (VTE) is a condition in which people have problems due to the formation of blood clots in their veins.

The study drug rivaroxaban is an approved treatment for VTE in children and adults in Japan. It is a blood thinner that prevents the blood from clotting by blocking a protein responsible for blood clotting.

Warfarin is another blood thinner that is available for VTE. In this study warfarin is the reference drug.

A previous study was carried out to learn about how well rivaroxaban works and how safe it is in children with VTE. However, to better understand the safety of this drug in children, more knowledge is needed about the use of rivaroxaban in the real world.

The main purpose of this study is to learn more about the occurrence of major bleeding in children taking rivaroxaban. Major bleeding can be bleeding within the skull, bleeding inside the eye, bleeding from an organ in the digestive system, or bleeding which requires being given blood from a donor.

In addition, this study will help learn more about the following in children with VTE:

* The occurrence of major bleeding during treatment with rivaroxaban and during treatment with warfarin
* The occurrence of bleeding of importance in children being treated with rivaroxaban and in children being treated with warfarin. Bleeding of importance in children can be: bleeding from the lung, blood in the kidney, heavy menstrual bleeding
* The occurrence of major bleeding and bleeding of importance in children who are taking drugs called anti platelet agents and NSAIDs to prevent blood clots at the same time as rivaroxaban, who are taking a drug that blocks the action of a protein called 'CYP3A4' at the same time as rivaroxaban, who have reduced kidney function, who have taken rivaroxaban for a long time, or who have taken other drugs by mouth to prevent blood clots before starting rivaroxaban
* The occurrence of repeated VTE on treatment with rivaroxaban and on treatment with warfarin The children with VTE in this study are already receiving rivaroxaban or warfarin treatment as part of their regular care from their doctors.

The data will come from an electronic health records database created by a company called Medical Data Vision. The data will be collected between January 2021 and June 2024.

Researchers will look at the health information from children less than 18 years of age with VTE in Japan who are prescribed treatment with rivaroxaban or warfarin during the study period.

In this study, only available data from routine care are collected. No visits or tests are required as part of this study

ELIGIBILITY:
Inclusion Criteria:At index date, which is the date of first prescription of rivaroxaban or of warfarin during the study period

* Age less than 18 years
* Diagnosis of VTE at any point before and including the index date
* Receiving a prescription/dispensation of rivaroxaban or warfarin

Exclusion Criteria:

* none

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with pediatric VTE treated with rivaroxaban or warfarin in real-world clinical practice in Japan between 01 January 2021 and 30 June 2024
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Incidence of major bleeding in participants treated with rivaroxaban | Retrospective analysis from January 2021 to June 2024
  Major bleeding is defined as composite of composite of intracranial hemorrhage, intraocular bleeding, upper gastrointestinal bleeding, lower gastrointestinal bleeding, bleeding requiring for blood transfusion
Clinical characteristics and demographics of participants with pediatric VTE treated with rivaroxaban | Retrospective analysis from January 2021 to June 2024
  Characteristics and demographics of participants will include e.g., age and gender, diagnosis and prior treatment, past medical history, concomitant diseases, and concomitant medication. They will be described.

SECONDARY OUTCOMES:
Incidence of major bleeding in participants treated with warfarin | Retrospective analysis from 01 January 2021 to 30 June 2024
  Major bleeding is defined as composite of composite of intracranial hemorrhage, intraocular bleeding, upper gastrointestinal bleeding, lower gastrointestinal bleeding, bleeding requiring for blood transfusion
Incidence of bleeding important in pediatrics in participants treated with rivaroxaban and treated with warfarin as reference | Retrospective analysis from 01 January 2021 to 30 June 2024
  Bleeding important in pediatrics is defined as composite of pulmonary hemorrhage, renal hemorrhage, hypermenorrhea
Incidence of major bleeding and bleeding important in pediatrics in participants treated with rivaroxaban and in special target patient groups | Retrospective analysis from 01 January 2021 to 30 June 2024
  target patient groups:
  * concomitant use with anti-platelet agents and NSAIDs
  * concomitant use with CYP3A4 inhibitors
  * impaired renal function
  * long term administration
  * other oral anti-coagulants administration prior to rivaroxaban

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Many facilities, Multiple Locations
  - Bayer, Osaka

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — https://clinicaltrials.bayer.com